CLINICAL TRIAL: NCT06559566
Title: Comparison of Two Methods Used to Asses Postoperative Intracranial Pressure in Patients Undergoing Intracranial Tumor Surgery
Brief Title: Evaluation of Postoperative Intracranial Pressure in Patients Undergoing Intracranial Tumor Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sezen Kumaş Solak (Other Government)
Collaborators: Bagcilar Training and Research Hospital (Other Government)
Responsible Party: Sponsor-Investigator, Sezen Kumaş Solak, SPONSOR INVESTIGATOR, Bagcilar Training and Research Hospital
Organization: Bagcilar Training and Research Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: BAGCILAR 3
Record Dates: First submitted 2024-07-31; First posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: INTRACRANIAL TUMOR; INTRACRANIAL PRESSURE; OPTIC NERVE
Keywords: OPTIC NERVE; INTRACRANIAL PRESSURE; INTRACRANIAL TUMOR; INTRACRANIAL TUMOR SURGERY; Intracranial Pressure Change
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ONSD measurement with USG (Active Comparator): After the ONSD measurement is made before anesthesia induction, general anesthesia will be given to each patient according to the institutional protocol. The ONSD measurements of the patients will be measured according to the T0, T1, T2, T3, T4, T5 time period by a person who has experience in using USG T0: Before anesthesia induction T1: First 5 minutes immediately after induction of anesthesia T2: At the end of the surgery before extubation /minute T3: Within the first hour/minute after extubation T4: 12 hours/minute after tumor resection T5. 24 hours/minute after tumor resection
  Interventions: Procedure: USG
- ONSD measurement with BCT (Active Comparator): In patients, USG and BCT correlation comparison is planned before the operation (T0), in the first hour after the end of post-operative surgery (T3) and at the 24th hour after post-operative surgery (T5).
  T0: ONSD measurement in pre-operative BCT T3: BCT ONSD measurement/minute within the first hour following the postoperative period T5: BCT ONSD measurement/minute 24 hours following the postoperative period The measurement of ONSD in BCT is; Eyeball diameter and optic nerve diameter measurements will be made on BCT transverse images at the optic nerve level and recorded.
  Interventions: Procedure: BCT

INTERVENTIONS:
Procedure: USG — The aim of this study is to measure the intracranial pressure of patients planned for brain tumor surgery by measuring the optic nerve sheath diameter (ONSD) under USG guidance and compare its correlation with the computed brain tomography.
  Other Names: ONSD measurement with USG
  Arms: ONSD measurement with USG
Procedure: BCT — The aim of this study is to measure the intracranial pressure of patients planned for brain tumor surgery by measuring the optic nerve sheath diameter (ONSD) under USG guidance and compare its correlation with the computed brain tomography.
  Other Names: ONSD measurement with BCT
  Arms: ONSD measurement with BCT

SUMMARY:
Ultrasonography(USG)-guided optic nerve sheath diameter measurement and its correlation with brain computed tomography in the evaluation of intracranial pressure in patients who underwent intracranial brain tumor surgery.

DETAILED DESCRIPTION:
Optic Nerve Sheath Diameter (ONSD) Measurement is a non-invasive diagnostic method used to detect increased intracranial pressure, and in general, ONSD measurement over 5 mm has been found to be associated with increased intracranial pressure.ONSD will be measured using an USG device within the specified time periods.

T0: Before anesthesia induction T1: First 5 minutes immediately after induction of anesthesia T2: At the end of the surgery before extubation /minute T3: Within the first hour/minute after extubation T4: 12 hours/minute after tumor resection T5. 24 hours/minute after tumor resection

ONSD measurement in brain computer tomography (BCT); Eyeball diameter and optic nerve diameter measurements will be made on BCT transverse images at the optic nerve level and recorded.In patients, USG and BCT correlation comparison is planned before the operation (T0), in the first hour after the end of post-operative surgery (T3) and at the 24th hour after post-operative surgery (T5).

T0: ONSD measurement in pre-operative Brain CT T3: BCT ONSD measurement/minute within the first hour following the postoperative period T5: BCT ONSD measurement/minute 24 hours following the postoperative period

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 -65 years
* Brain malignant neoplasm tumor
* Brain benign neoplasm supratentorial
* Brain benign neoplasm infratentorial information

Exclusion Criteria:

* Patients who cannot provide adequate image quality in ocular ultrasonography
* Who are unconscious or have a Glasgow coma scale of less than 15
* Pseudotumor cerebri
* Optic nerve arachnoid cyst
* Patients with open injuries involving the eyelid and surrounding area
* Optic nerve malignant neoplasm
* Injury of the optic nerve and its pathways
* Systemic Lupus Erythematosis,
* Scleroderma
* Multiple Sclerosis, sarcoidosis
* Thyrotoxicosis (hyperthyroidism)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-09-15 (Estimated); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
intracranial pressure | T0: Before anesthesia induction T1: peroperative5. minutes T2: At the end of the surgery 6.hours T3:after extubation 1 hours T4: postoperative 12.hours T5. postoperative 24.hours
  To compare the optic nerve diameter measurement ,USG and BBT values used to measure intracranial pressure in patients with brain tumor surgery

SECONDARY OUTCOMES:
Heart Rate | T0: Before anesthesia induction T1: preoperative 5.minutes T2: At the end of the surgery 6.hoursT3:after extubation 1 hours T4: postoperative 12.hours T5. postoperative 24.hours
  To compare the heart rate measurement
Blood pressure | T0: Before anesthesia induction T1: preoperative 5.minutes T2: At the end of the surgery 6.hours T3 extubation 1 hours T4: postoperative 12.hours T5. postoperative 24.hours
  To compare the blood pressure measurement

CONTACTS AND LOCATIONS:
Overall Officials: SEZEN KUMAS SOLAK, MD, Principal Investigator — Bagcılar Training Research Hospital

IPD SHARING:
Plan to Share IPD: No
The investigators will not share individual patient data

REFERENCES:
- [Background] Stevens RRF, Gommer ED, Aries MJH, Ertl M, Mess WH, Huberts W, Delhaas T. Optic nerve sheath diameter assessment by neurosonology: A review of methodologic discrepancies. J Neuroimaging. 2021 Sep;31(5):814-825. doi: 10.1111/jon.12906. Epub 2021 Jul 16. PMID 34270144
- [Background] Raffiz M, Abdullah JM. Optic nerve sheath diameter measurement: a means of detecting raised ICP in adult traumatic and non-traumatic neurosurgical patients. Am J Emerg Med. 2017 Jan;35(1):150-153. doi: 10.1016/j.ajem.2016.09.044. Epub 2016 Sep 23. PMID 27852525
- [Background] Xu J, Song Y, Shah Nayaz BM, Shi W, Zhao Y, Liu Y, Wu S, Li Z, Sun Y, Zhao Y, Yu W, Wang X. Optic Nerve Sheath Diameter Sonography for the Diagnosis of Intracranial Hypertension in Traumatic Brain Injury: A Systematic Review and Meta-Analysis. World Neurosurg. 2024 Feb;182:136-143. doi: 10.1016/j.wneu.2023.11.016. Epub 2023 Nov 10. PMID 37951461